CLINICAL TRIAL: NCT00272519
Title: Life Skills Intervention for Young Adolescents Perinatally Infected With HIV and Their Caregivers
Brief Title: Life Skills Intervention for Adolescents Perinatally Infected With HIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); National Institute of Mental Health (NIMH) (NIH); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: ATN 045b
Record Dates: First submitted 2006-01-03; First posted 2006-01-06 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2016-02

CONDITIONS: HIV Infections
Keywords: HIV; AIDS; Adolescent; HIV Positive
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; HIV Seropositivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Adolescent/caregiver dyads (Experimental): Eight to ten adolescent/caregiver dyads
  Interventions: Behavioral: Life Skills Intervention

INTERVENTIONS:
Behavioral: Life Skills Intervention — Developed to promote life skills among young adolescents perinatally infected with HIV
  Other Names: No other names.

SUMMARY:
The life skills intervention model is designed to help adolescents promote their physical and mental health through cognitive and behavioral techniques (e.g., problem solving, coping, and communication skills) designed to help them achieve social and personal competencies used to manage various life challenges.

DETAILED DESCRIPTION:
One of the salient advantages of this intervention model is that it has been developed and implemented in several studies with adolescents. However, data concerning the effects of this model are much less extensive with adolescents perinatally infected with HIV. The proposed study is designed to address this gap in knowledge by conducting a pilot intervention tailoring the life skills intervention to the needs of young adolescents, perinatally infected with HIV, and to their primary caregivers. Given the emphasis on peer group interaction, the proposed intervention model also has the potential to reduce some of the social isolation imposed by the experiences related to HIV infection by creating opportunities for adolescents to interact with others who are managing comparable stressors and treatment regimens.

ELIGIBILITY:
Inclusion Criteria:

* Clinically-identified HIV-1 infected participants 11-14 years of age and their primary caregivers.
* HIV status has been disclosed to the adolescent.
* Caregiver is the legal guardian of the adolescent as indicated by the medical team.
* Adolescent lives with the caregiver
* Adolescent and caregiver speak and understand English.

Exclusion Criteria:

* Caregiver consent or permission denied or adolescent does not assent.
* Adolescent diagnosed as mentally retarded as previously reported or confirmed through chart review.
* Adolescent and/or caregiver too medically fragile. Medically fragile is functionally defined as being physically unable to attend the group.

Ages: 11 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2006-06; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Implement and evaluate the feasibility and acceptability of a modified life skills intervention | 1 year
  To implement and evaluate the feasibility and acceptability of a modified life skills intervention for young adolescents with perinatally acquired HIV infection and their primary caregivers.

SECONDARY OUTCOMES:
Evaluate the feasibility and acceptability of an assessment battery | 1 year
  To evaluate the feasibility and acceptability of an assessment battery with young adolescents with perinatally acquired HIV infection and their primary caregivers when implemented at baseline, post-intervention and 4-month follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Ahna Pai, Ph.D, Study Chair — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Website for the Adolescent Trials Network for HIV/AIDS Interventions — http://www.atnonline.org